CLINICAL TRIAL: NCT07380607
Title: Sensitivity of Diaphragmatic Ultrasonography in Detecting Double Triggering Asynchrony in Mechanically Ventilated ICU Patients.
Brief Title: Double Triggering Asynchrony in Mechanically Ventilated Patients.
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: MD.24.03.838.R1
Record Dates: First submitted 2026-01-17; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Patient-Ventilator Asynchrony Double Triggering Asynchrony Critical Illness
Keywords: double triggering ventilator asynchrony mechanical ventilation ICU diaphragmatic ultrasound cross-sectional study

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Double Triggering Cohort: 28mechanically ventilated ICU patients identified with double triggering asynchrony

SUMMARY:
This observational study examined double triggering asynchrony in28ICU patients on mechanical ventilation. Researchers collected data on patient characteristics, health conditions, and outcomes to understand how this problem affects critically ill patients. Findings may help improve ventilator care in intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* Adult ICU patients aged ≥18 years receiving invasive mechanical ventilation
* Documented double triggering asynchrony on ventilator waveform analysis.

Exclusion Criteria:

* Patients with contraindications to diaphragmatic ultrasound, including thoracic or abdominal surgery.
* Patients with known diseases affecting diaphragmatic function, such as Duchenne muscular dystrophy (DMD) or myasthenia gravis (MG).
* Patients with advanced chronic liver disease (Child-Pugh class C)
* Patients with chronic increased intra-abdominal pressure.
* Patients with moderate to massive pleural effusion.
* Patient or legal guardian refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years) admitted to medical/surgical ICU at Specialized Medical Hospital, Mansoura University, receiving invasive mechanical ventilation with documented double triggering asynchrony on ventilator waveform analysis.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-11-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity of diaphragmatic ultrasound for detection of double triggering asynchrony | During ICU admission, at the time of double triggering detection by ventilator graph interpretation
  Proportion of double triggering asynchrony events correctly identified by diaphragmatic ultrasound compared with ventilator waveform analysis as the reference standard

CONTACTS AND LOCATIONS:
Locations (1):
- Specialised Medical Hospital - ICU, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No